CLINICAL TRIAL: NCT04233905
Title: A Psychometric Questionnaire Study With a Control Group Design of Children and Young People With Selective Mutism, as Well as on Adults Who Suffered Selective Mutism Earlier in Life
Brief Title: Factors Influencing Selective Mutism
Status: Completed | Type: Observational
Sponsor: Susanne Walitza (Other)
Responsible Party: Sponsor-Investigator, Susanne Walitza, Head of the Department of Child and Adolescent Psychiatry, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Other Study IDs: KJPP 2017-00679
Record Dates: First submitted 2019-12-05; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Selective Mutism
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- mute children: mute children and their mothers
  Interventions: Behavioral: Psychometric questionnaire study
- healthy children: healthy children control group
  Interventions: Behavioral: Psychometric questionnaire study
- mute adults: formerly mute adults
  Interventions: Behavioral: Psychometric questionnaire study
- healthy adults: healthy adults control group
  Interventions: Behavioral: Psychometric questionnaire study

INTERVENTIONS:
Behavioral: Psychometric questionnaire study — Four groups participate in the psychometric questionnaire study. A group of mute children and their mothers (EG:A), as well as a normal, healthy control group (KG:A) with roughly the same age and sex characteristics fill out one-time questionnaires about current daily life experiences. In addition, another group of formerly mute adults (EG:B) as well as a comparable age/sex normal control group will be retrospectively questioned using the same specifically tailored questionnaire.

SUMMARY:
The study's goal is to check and verify basic assumptions of a new selective mutism developmental model from Melfsen and Walitza through standardized and routinely used patient questionnaires. The primary emphasis is the question of a connection between selective mutism and high sensitivity, dissociation, emotional regulation, family structure, social anxiety and self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people from 8-18 years of age who fulfill the international classification of diseases tenth edition (ICD-10) for selective mutism
* Adults who suffered selective mutism when they were children or adolescents
* All study participants or their legal representative have given written permission for their experiences to be documented in the study.

Exclusion Criteria:

* Temporary mutism, e.g. from emotional disturbances or separation anxiety (F93.0), or depression
* Profound developmental disturbances (F84.2) like early childhood autism (F84.0), atypical autism (F84.1), Rett Syndrome (F84.2), alternative disintegrative childhood disturbances (F84.3), hyperactivity disturbance with decrease of intelligence and movement stereotypes (F84.5), or Asperger's Syndrome.
* Schizophrenia (F20)
* Profound mental retardation
* Delineated development disturbances of speech and language (F80)
* Organic brain disease with loss of language or disturbance of speech development

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample consist of pupils with selective mutism aged 8 to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Symptoms severity of selective mutism | 24 months
  The parent report "Selective Mutism Questionnaire (SMQ)" is a 17-item parent-rating measure designed to assess the severity of selective mutism. The test uses a 4-point scale to rate the frequency of the child's speaking behaviour in school (6 items), home/family (6 items) and public settings outside school (5 items) from 0 (never) to 3 (always) each, with a total score of 51. Higher score means a worse outcome.
High sensitivity | 24 months
  The "Highly Sensitive Person Scale" (HSP) is a self-report questionnaire with 27 items to be answered on a seven-point Likert scale (from 1 "not at all" to 7 "absolutely"). The total score divided by item number ranges from 0 to 7. Higher score means a worse outcome.
Family relation structure | 24 months
  The "Parent-Image-Questionnaire for Children and Adolescents (EBF-KJ)" is a self-reporting questionnaire for children and adolescents to record the family relationship structure with 36 items on a five-point Likert scale from 0 (never) to 4 (always). Higher score means a stronger characteristic.
Emotion regulation | 24 months
  Emotion regulation is measured using the German questionnaire "Fragebogen zur Erhebung der Emotionsregulation bei Kindern und Jugendlichen (FEEL-KJ). It is a multi-dimensional tool for the emotion-specific detection of emotion regulation strategies. It measures fear, sadness and anger. Adaptive strategies include problem-oriented behavior, dispersion, mood elevation, acceptance, forgetting, revaluation and cognitive problem solving. Maladaptive strategies include abandonment, aggressive behavior, withdrawal, self-devaluation and perseveration. A total of 90 items is to be rated on the basis of a five-level rating scale with regard to their frequency. Higher scores mean more adaptive or maladaptive strategies.
Symptoms of selective mutism | 24 months
  Symptom severity is assessed by using the "Checklist for speaking behaviour, parent report" (CheckS). It assesses the communicative burden of various socially interactive situations for children suffering from selective mutism on a five-point scale (from 0 = "never" to 4 = "always"). A distinction is made between different contexts, namely the persons to be spoken to, the type of communication, the length of the spoken answers, the conversational situations, the contents of the conversation, the places and surroundings, the expectations of those present and the unpredictability of contexts. The total score ranges from 0 to 4.Higher score means a worse outcome.
Dissociation | 24 months
  The German translation of the "Child Dissociative Checklist" (CDC) is a parent report of 20 items using a three-point Likert scale (0 = "very true", 1 ="somewhat true", 2 ="not true"). Parents are asked to report dissociative behavioural problems of their child within the past 12 months. Higher score means a worse outcome.
Dissociation | 24 months
  The children and adolescents completed the "Self-Perception Questionnaire for Children and Adolescents" (A-DES) to assess dissociative symptoms. 30 items are to be assessed on an 11-point rating scale (from 0 = "never" to 10 = "always") in terms of their frequency. Higher score means a worse outcome.
Social anxiety | 24 months
  The German version of the "Social phobia and anxiety inventory for children (SPAIK) is used to asses social anxiety in children and adolescents. The questionnaire consists of 26 situations assessing somatic, cognitive and behavioural aspects of social anxiety. They measure characteristic aspects of social anxiety on a three-point Likert scale (from 0 = "never or seldom" to 3 = "most of the time or always") with a total score of 52. Higher score means a worse outcome.
Self-esteem | 24 months
  The "List of statements on self-esteem for children and adolescents" (ALS) uses the same 18 items to differentiate the self-esteem of children and adolescents in three areas: family, school and leisure. Higher score means a stronger self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Walitza, Prof. Dr. med. Dipl.-Psych., Principal Investigator — Sponsor-Investigator
Locations (1):
- Psychiatric University Clinics, Department of Child and Adolescent Psychiatry, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Melfsen S, Jans T, Romanos M, Walitza S. Emotion regulation in selective mutism: A comparison group study in children and adolescents with selective mutism. J Psychiatr Res. 2022 Jul;151:710-715. doi: 10.1016/j.jpsychires.2022.05.040. Epub 2022 May 24. PMID 35690008
- [Derived] Melfsen S, Romanos M, Jans T, Walitza S. Betrayed by the nervous system: a comparison group study to investigate the 'unsafe world' model of selective mutism. J Neural Transm (Vienna). 2021 Sep;128(9):1433-1443. doi: 10.1007/s00702-021-02404-1. Epub 2021 Aug 14. PMID 34390394